CLINICAL TRIAL: NCT00603096
Title: Interest of Using Nocturnal Polysomnography for Non-Invasive Ventilation (NIV) Settings' Optimization in Obesity-Hypoventilation Syndrome (OHS)
Brief Title: Use of Polysomnography for Non-Invasive Ventilation Settings' Optimization
Acronym: NIV-OHS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tyco Healthcare Group (Industry)
Responsible Party: EMEA Clinical Affairs Director, tyco Healthcare Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38/2006/2; Ethics Comittee ref.06-TYCO-1
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2008-01

CONDITIONS: Obesity-Hypoventilation Syndrome (OHS)
MeSH Terms: conditions — Obesity Hypoventilation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): patients will benefit from a complete polysomnography under NIV
  Interventions: Device: GoodKnight 425ST - Mallinckrodt DF, Tyco Healthcare
- 2 (Active Comparator): settings will be adjusted using only nocturnal oxygen SaO2 and PaCO2 at awakening whereas
  Interventions: Device: GoodKnight 425ST - Mallinckrodt DF, Tyco Healthcare

INTERVENTIONS:
Device: GoodKnight 425ST - Mallinckrodt DF, Tyco Healthcare — The aim of this randomized controlled trial is comparing the improvement of diurnal PaCO2 in OHS patients after one month of NIV treatment depending upon the tools used for adjusting settings. In one arm settings will be adjusted using only nocturnal oxygen SaO2 and PaCO2 at awakening whereas in the other arm patients will benefit from a complete polysomnography under NIV.

SUMMARY:
The aim of this randomized controlled trial is comparing the improvement of diurnal PaCO2 in OHS patients after one month of NIV treatment depending upon the tools used for adjusting settings. In one arm settings will be adjusted using only nocturnal oxygen SaO2 and PaCO2 at awakening whereas in the other arm patients will benefit from a complete polysomnography under NIV.

DETAILED DESCRIPTION:
Initiation of NIV treatment implies technical adjustments (choice of mask and ventilator), but also patient education by the nurses and medical staff. The settings are generally adjusted during the daytime in awake patients. The appropriateness of these settings is generally not optimal during sleep as many respiratory events (hypopnoea, apnea, leaks, desynchronization, and glottic closure) may occur under NIV then reducing the effectiveness of treatment. These nocturnal abnormalities are routinely evaluated by measuring their consequences, i.e. oxygen desaturation and the level of PaCO2 after wake up. Some teams are now proposing to better characterize what happens when using NIV during sleep using polysomnography (PSG). The precise characterization of residual events under treatment may allow optimizing ventilator settings.

ELIGIBILITY:
Inclusion Criteria:

* Patient male or female, aged 20 to 75 years
* Patient with a OHS in stable condition, with a BMI> 32 kg/m2 and a PaCO2> 6 kPa in diurnal spontaneous breathing without other cause of alveolar hypoventilation
* Patient affiliated to a social security insurance
* Having given its written informed consent to participate to the study

Exclusion Criteria:

* Patients with inherent chronic obstructive pulmonary disease (COPD) with FEV1 on Forced Vital Capacity (FVC) ratio less than 70%
* Patients suffering from heart failure with periodic breathing
* Associated Neurological Diseases, evolving rapidly, leading to a dependency in daily activities
* Unbalanced Psychiatric Diseases
* Patients with a respiratory decompensation the month preceding the study
* Patients not autonomous in the use of the NIV
* Pacemaker patients, constituting a contraindication to magnetic stimulation
* Sensitive subjects, in accordance with article L 1121-6 of the French Public Health Code
* Patients with long term by steroids or other anti-inflammatory drugs

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2006-06; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Diurnal PaCO2 | June 2008

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis pepin, Pr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Laboratoire d'Explorations Fonctionnelles Cardio-Respiratoires - CHU Grenoble, Grenoble, Cedex 9, France

REFERENCES:
- [Derived] Borel JC, Tamisier R, Gonzalez-Bermejo J, Baguet JP, Monneret D, Arnol N, Roux-Lombard P, Wuyam B, Levy P, Pepin JL. Noninvasive ventilation in mild obesity hypoventilation syndrome: a randomized controlled trial. Chest. 2012 Mar;141(3):692-702. doi: 10.1378/chest.10-2531. Epub 2011 Sep 1. PMID 21885724
- [Derived] Borel JC, Roux-Lombard P, Tamisier R, Arnaud C, Monneret D, Arnol N, Baguet JP, Levy P, Pepin JL. Endothelial dysfunction and specific inflammation in obesity hypoventilation syndrome. PLoS One. 2009 Aug 24;4(8):e6733. doi: 10.1371/journal.pone.0006733. PMID 19701463